CLINICAL TRIAL: NCT02796014
Title: Assessment of Dermatologic Family Impact Scale in the Parents of Children With Psoriasis, and Comparison of This Scale With the Children's Dermatology Life Quality Index and Disease Severity
Brief Title: Assessment of Dermatologic Family Impact Scale in the Parents of Children With Psoriasis
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government); Haseki Training and Research Hospital (Other); Haydarpasa Numune Training and Research Hospital (Other); Istanbul Training and Research Hospital (Other Government); Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other); Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, burak tekin, Dr, M.D., Istanbul Medeniyet University
Other Study IDs: 2016/0118
Record Dates: First submitted 2016-06-07; First posted 2016-06-10 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Psoriasis; Quality of Life
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Dermatological Diseases Family Impact Scale (DeFIS) was developed to assess different aspects of health-related quality of life in the relatives of the patients with various skin diseases. The preliminary validation of this instrument was performed for the Turkish population. In the pilot study, this 15-item-questionnaire was shown to be easy to complete and score, and reliably help to evaluate the family members' quality of life.

Psoriasis is a chronic disease which can be expected to have a significant impact on the quality of life of the patients and parents/family members alike. In line with this assumption, previous studies demonstrated that psoriasis psychosocially affects not only the patients, but also their close relatives. The psoriasis family index has been developed in an effort to objectively measure the health-related quality of life of the family members of patients with psoriasis. Nevertheless, data regarding the health-related quality of life of the parents of pediatric patients with psoriasis in the Turkish population are relatively scarce.

In study, the investigators primarily aim to utilize DeFIS to assess the impact of childhood psoriasis on the quality of life of the patients' parents. Further, the investigators attempt to investigate the relation between the quality of life of the patients and their parents, and reveal disease characteristics which might influence the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients diagnosed with psoriasis by the dermatologists within the study period

Exclusion Criteria:

* Patients with an equivocal diagnosis
* Parents unable to complete the questionnaire
* Patients with a serious medical disorder or in an emergency condition

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients clinically (andif necessary histopathologically) diagnosed with psoriasis < 18 years of age
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2016-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Assessment of the impact of childhood psoriasis on the parents of the patients using the Dermatological Diseases Family Impact Scale | 6 months

SECONDARY OUTCOMES:
Comparison of the quality of life of the parents (as evaluated using the Dermatological Diseases Family Impact Scale) with the quality of life of the patients (as assessed using the Children's Dermatology Life Quality Index) | 6 months
Delineating disease characteristics which influence the patients' and/or their parents' health-related quality of life | 6 months
  Disease characteristics such as age of onset, disease subtype, psoriasis area and severity index and scalp involvement will be recorded. The impact of these parameters on quality of life will be assessed using statistical methods.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Tekin, M.D., Principal Investigator — Istanbul Medeniyet University Goztepe Research and Training Hospital Department of Dermatology
Locations (7):
- Turkey (Türkiye) (7):
  - Istanbul Medeniyet University Goztepe Research and Training Hospital, Istanbul, Kadikoy
  - Bakirkoy Dr. Sadi Konuk Research and Training Hospital, Istanbul
  - Haseki Training and Research Hospital, Istanbul
  - Haydarpasa Numune Training and Research Hospital, Istanbul
  - Istanbul Training and Research Hospital, Istanbul
  - Okmeydani Training and Research Hospital, Istanbul
  - Sisli Etfal Training & Research Hospital, Istanbul

REFERENCES:
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- [Background] Gurel MS, Yanik M, Simsek Z, Kati M, Karaman A. Quality of life instrument for Turkish people with skin diseases. Int J Dermatol. 2005 Nov;44(11):933-8. doi: 10.1111/j.1365-4632.2004.02225.x. PMID 16336527
- [Background] Lewis-Jones MS, Finlay AY. The Children's Dermatology Life Quality Index (CDLQI): initial validation and practical use. Br J Dermatol. 1995 Jun;132(6):942-9. doi: 10.1111/j.1365-2133.1995.tb16953.x. PMID 7662573
- [Background] Basra MK, Sue-Ho R, Finlay AY. The Family Dermatology Life Quality Index: measuring the secondary impact of skin disease. Br J Dermatol. 2007 Mar;156(3):528-38. doi: 10.1111/j.1365-2133.2006.07617.x. PMID 17300244
- [Background] Eghlileb AM, Basra MK, Finlay AY. The psoriasis family index: preliminary results of validation of a quality of life instrument for family members of patients with psoriasis. Dermatology. 2009;219(1):63-70. doi: 10.1159/000209234. Epub 2009 Mar 13. PMID 19295185
- [Background] Tadros A, Vergou T, Stratigos AJ, Tzavara C, Hletsos M, Katsambas A, Antoniou C. Psoriasis: is it the tip of the iceberg for the quality of life of patients and their families? J Eur Acad Dermatol Venereol. 2011 Nov;25(11):1282-7. doi: 10.1111/j.1468-3083.2010.03965.x. Epub 2011 Jan 17. PMID 21241373
- [Background] Ganemo A, Wahlgren CF, Svensson A. Quality of life and clinical features in Swedish children with psoriasis. Pediatr Dermatol. 2011 Jul-Aug;28(4):375-9. doi: 10.1111/j.1525-1470.2010.01292.x. Epub 2011 Jul 8. PMID 21736605
- See also: Development and preliminary validation of the dermatological family impact scale — http://journal.turkderm.org.tr/jvi.aspx?pdir=turkderm&plng=tur&un=TURKDERM-27167